CLINICAL TRIAL: NCT05311423
Title: The Prevalence of Genital Tuberculosis and the Impact on Reproductive Outcomes in Infertile Women: a National Multicenter Prospective Cohort Study
Brief Title: The Prevalence and Reproductive Outcome of Infertile Women With Genital Tuberculosis
Acronym: TB-PRIME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai First Maternity and Infant Hospital (Other); General Hospital of Ningxia Medical University (Other); Tang-Du Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The First Affiliated Hospital of Zhengzhou University (Other); The 924th Hospital of Joint Logistics Support Force of Chinese People's Liberation (Unknown); Shenzhen Zhongshan Urology Hospita (Unknown); Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other); Jiangxi Maternal and Child Health Hospital (Other); The First People's Hospital of Yunnan (Other); Tongji Hospital (Other); The Second Hospital of Hebei Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, director of department of infectious diseases, Huashan Hospital
Other Study IDs: KY2021-840
Record Dates: First submitted 2022-01-21; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Infertility, Female; Genital Tuberculoses, Female
MeSH Terms: conditions — Infertility, Female; Tuberculosis, Female Genital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-TB Group: QuantiFERON-TB test (QFT) negative, continue assisted reproductive treatment
  Interventions: Diagnostic Test: QuantiFERON-TB test & endometrial pathology & endometrial tissue GeneXpert Ultra
- Latent tuberculosis infection Group: QFT positive. Excluded active pulmonary tuberculosis, patients have negative endometrial histopathology, acid-fast bacilli (AFB) microscopy, Mycobacterium tuberculosis (Mtb) culture, or GeneXpert MTB/RIF Ultra test results. Then assisted reproductive treatment can be continued, but follow-up for tuberculosis-related symptoms is required
  Interventions: Diagnostic Test: QuantiFERON-TB test & endometrial pathology & endometrial tissue GeneXpert Ultra
- Subclinical genital tuberculosis Group: QFT positive. Excluded active pulmonary tuberculosis, patients have negative endometrial histopathology, AFB microscopy, Mtb culture, but GeneXpert MTB/RIF Ultra positive test results. They are recommended to receive 6-month first-line standard anti-tuberculosis treatment (ATT) regimen
  Interventions: Diagnostic Test: QuantiFERON-TB test & endometrial pathology & endometrial tissue GeneXpert Ultra
- Female genital tuberculosis Group: QFT positive. Excluded active pulmonary tuberculosis, regardless of GeneXpert MTB/RIF Ultra results, at least one of these test results, including endometrial histopathologiy, AFB microscopy, Mtb culture is positive, they will receive 6-month ATT
  Interventions: Diagnostic Test: QuantiFERON-TB test & endometrial pathology & endometrial tissue GeneXpert Ultra

INTERVENTIONS:
Diagnostic Test: QuantiFERON-TB test & endometrial pathology & endometrial tissue GeneXpert Ultra — Endometrial biopsy is required to diagnose LTBI, SGTB and FGTB, which is an invasive operation and increases patients' economic burden. A screening method has been established that uses the interferon gamma release test as the primary screening test, and those who are positive undergo endometrial biopsy. Therefore, this project will use QFT to screen participants with Mtb infection, and further endometrium biopsy will be performed for QFT positive patients to diagnose LTBI, FGTB and SGTB. For participants with negative results for all diagnostic tests but QFT (defined as LTBI), close follow-up is necessary according to WHO guidelines.

SUMMARY:
Female genital tuberculosis infection (FGTB) is an important cause of female infertility in TB-endemic areas. The pregnancy rate of assisted reproductive treatment (ART) in the infertile women with FGTB is still unsatisfied even after receiving standard anti-tuberculosis treatment. Moreover, recent years have witnessed an alarming increase in reports of FGTB-related maternal and neonatal complications after fertility treatments. These underscore that timely detection and treatment of FGTB before ART hold benefit for the mother and child.

DETAILED DESCRIPTION:
This project aims to recruit infertile female with high risk of tuberculosis infecton who need assisted reproductive treatment in multiple reproductive centers. The infertility-related medical history and laboratory examination results were recorded according to clinical routine, and other essential information such as tuberculosis symptoms, tuberculosis-related history and other health conditions were also recorded, and the pregnancy outcomes of these patients were followed up.

According to the results of clinical screening, they were divided into four cohorts: non-tuberculosis (non-TB) group, latent tuberculosis infection (LTBI) group, subclinical genital tuberculosis infection (SGTB) group and female genital tuberculosis infection (FGTB) group.

Non-TB group: QuantiFERON-TB test (QFT) negative, continue assisted reproductive treatment; LTBI group: QFT positive. Excluded active pulmonary tuberculosis, patients have negative endometrial histopathology, acid-fast bacilli (AFB) microscopy, Mycobacterium tuberculosis (Mtb) culture, or GeneXpert MTB/RIF Ultra test results. Then assisted reproductive treatment can be continued, but follow-up for tuberculosis-related symptoms is required; SGTB group: QFT positive. Excluded active pulmonary tuberculosis, patients have negative endometrial histopathology, AFB microscopy, Mtb culture, but GeneXpert MTB/RIF Ultra positive test results. They are recommended to receive 6-month first-line standard anti-tuberculosis treatment (ATT) regimen; FGTB group: QFT positive. Excluded active pulmonary tuberculosis, regardless of GeneXpert MTB/RIF Ultra results, at least one of these test results, including endometrial histopathologiy, AFB microscopy, Mtb culture is positive, they will receive 6-month ATT.

Patients diagnosed with SGTB and FGTB will receive 6-month first-line standard ATT before ART, and follow up their anti-tuberculosis drug-related adverse reactions (TB-ARs) according to clinical routine to prevent the occurrence of grade 3-4 adverse drug reactions.

All cohorts will be followed up for pregnancy outcomes after entering the assisted reproduction cycle, and the pregnancy outcomes of all subjects after the first assisted reproduction after enrollment were recorded. Follow-up nodes included the 2nd, 4th, 10th weeks and 37th weeks of gestation. Follow-up content includes pregnancy status. Follow-up subjects will be terminated when adverse pregnancy outcomes such as ectopic pregnancy and miscarriage occurred; follow-up of pregnant participants will be extended to 2 weeks postpartum. Participants from the SGTB or FGTB group achieve pregnant naturally after drug withdrawal, the follow-up of the natural pregnancy outcome will be started as well.

ELIGIBILITY:
Inclusion Criteria:

* 1) Female, aged ≥20 years and <43 years old;
* 2) In line with conventional assisted reproduction indications;
* 3) Meet any of the following:

  1. with tuberculosis infection history;
  2. with a history of close contact to tuberculosis patients;
  3. exact positive IGRA results in the past or chest imaging indicated a past history of pulmonary tuberculosis;
  4. suspected symptoms of tuberculosis, including fever, night sweats, fatigue, cough and sputum;
  5. suspected symptoms of genital tuberculosis, including lower abdominal pain, abnormal menstruation, fallopian tube stenosis, obstruction, thickening, beading changes, uterine cavity adhesions, deformation, pelvic adhesions, etc.;
* 4) Voluntarily join the study and sign the informed consent

Exclusion Criteria:

* 1) Co-infection with HIV;
* 2) Chromosomal abnormalities;
* 3) suspected genital tuberculosis infection symptoms (participants meet inclusion criteria 3)e in Inclusion Criteria) known to be caused only by factors part from tuberculosis, such as endocrine factors, history of ectopic pregnancy, history of uterine curettage, chronic pelvic inflammatory disease, endometriosis, malignant tumors, etc.;
* 4) There are other serious physical or mental illnesses that are not suitable for selection;
* 5) Participate in other clinical studies that would affect this study at the same time.

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile female patients with high risk factors for tuberculosis infection who intend to undergo assisted reproduction
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate of ART | 2 years
  the number of participants with gestational sacs seen by ultrasound examination 4-6 weeks after transplantation/the number of embryo transfer cycles in this group
Continued pregnancy rate of ART | 2 years
  the number of patients whose pregnancy was confirmed by repeat ultrasonography at 10th week of gestation/the number of embryo transfer cycles in this group
Prevalence of SGTB among infertile women | 6 months
  the number of SGTB participants/the total number of this project

SECONDARY OUTCOMES:
Prevalence of FGTB/LTBI among infertile women | 2 years
  the number of each group/the total number of this project
Abortion rate | 2 years
  number of abortions/number of clinical pregnancy in non-TB or LTBI or SGTB or FGTB group
Ectopic pregnancy rate | 2 years
  number of ectopic pregnancy/number of clinical pregnancy in non-TB or LTBI or SGTB or FGTB group
Preterm birth rate | 2 years
  the number of premature births/the number of clinical pregnancy in non-TB or LTBI or SGTB or FGTB group
Live birth rate | 2 years
  the number of live births/the number of clinical pregnancy in non-TB or LTBI or SGTB or FGTB group
Maternal mortality rate | 2 years
  the number of maternal mortality/the number of clinical pregnancy in non-TB or LTBI or SGTB or FGTB group
Neonatal mortality rate | 2 years
  the number of neonatal mortality/the number of clinical pregnancy in non-TB or LTBI or SGTB or FGTB group
Spontaneous pregnancy rate | 2 years
  number of Spontaneous pregnancy/number of subjects completed ATT in FGTB/SGTB group
The incidence of grade 3-4 adverse events | 2 years
  the number of patients with grade 3-4 adverse events during anti-tuberculosis treatment / the total number of in FGTB/SGTB group
The rate of drug discontinuation due to adverse drug reactions | 2 years
  the number of patients who discontinued in anti-tuberculosis treatment due to adverse drug reactions / the total number of patients with adverse reactions in FGTB/SGTB group
Treatment completion rate | 2 years
  number of patients who completed anti-tuberculosis treatment / total number of patients in this group × 100%
Incidence of active tuberculosis of LTBI group during 1 year after enrollment | 1 year
  the number of subjects who develop to active tuberculosis during 1 year after enrollment/the number of subjects of LTBI group

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality, China